CLINICAL TRIAL: NCT05423353
Title: Comparative Effects of Paraffin Bath Therapy and Extracorporeal Shock Wave Therapy on Pain and Hand Functions in Patients With De Quervain Tenosynovitis
Brief Title: Comparative Effects of Paraffin Bath Therapy and ESWT in Patients With De Quervain Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Van YYÜ School of Medicine
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: De Quervain Disease
MeSH Terms: conditions — De Quervain Disease | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin Bath Therapy (Active Comparator): Paraffin bath therapy is a physical therapy method that can create a temperature increase of 7.5 °C in the joint capsule and 4.5 °C in the muscle.
  Interventions: Device: Paraffin Bath Therapy
- Extracorporeal Shock Wave Therapy (Active Comparator): Extracorporeal shock wave therapy (ESWT) is a noninvasive treatment that involves delivery of shock waves to injured soft tissue to reduce pain and promote healing.
  Interventions: Device: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Paraffin Bath Therapy — Device named 'Fizyowax 1300' (Fizyomed, Turkey).
  Arms: Paraffin Bath Therapy
Device: Extracorporeal Shock Wave Therapy — Device named 'Elettronica Pagani,Italy' and will be used with radial probe.
  Arms: Extracorporeal Shock Wave Therapy

SUMMARY:
There is no study in the literature comparing both paraffin bath therapy and Extracorporeal Shock Wave Therapy (ESWT) in the treatment of patients with De Quervain Tenosynovitis. The aim of this study is performing this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Meeting De Quervain diagnostic criteria
* Not having applied any physical therapy modality to the hand-wrist in the last 1 month
* Not using pain medication in the last 1 month,
* Not using local anesthetics or steroid injections on the hand-wrist in the last 3 months
* Have received written consent to participate in the study, and have come to the last control at the 6th week.

Exclusion Criteria:

* Neurological diseases (especially neuropathies),
* Malignancy,
* Rheumatological diseases
* Pregnancy
* History of hand/wrist fracture or surgery
* Hand/wrist trauma in the last 1 month
* Coagulation disorder diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | at baseline (before the treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Visual Analogue Scale (VAS) | 2 weeks after baseline (at the end of treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Visual Analogue Scale (VAS) | 6 weeks after baseline (one month after the end of treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Duruöz Hand Index (DHI) | at baseline (before the treatment)
  Duruöz Hand Index (DHI) is a functional disability scale that can be used successfully to assess the functional disability with different hand arthropathies. It consists of 18 items that evaluate hand and wrist activities. The answers are evaluated on a 6-level (0-5) Likert scale and the total score ranges from 0 to 90.
Duruöz Hand Index (DHI) | 2 weeks after baseline (at the end of treatment)
  Duruöz Hand Index (DHI) is a functional disability scale that can be used successfully to assess the functional disability with different hand arthropathies. It consists of 18 items that evaluate hand and wrist activities. The answers are evaluated on a 6-level (0-5) Likert scale and the total score ranges from 0 to 90.
Duruöz Hand Index (DHI) | 6 weeks after baseline (one month after the end of treatment)
  Duruöz Hand Index (DHI) is a functional disability scale that can be used successfully to assess the functional disability with different hand arthropathies. It consists of 18 items that evaluate hand and wrist activities. The answers are evaluated on a 6-level (0-5) Likert scale and the total score ranges from 0 to 90.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No